CLINICAL TRIAL: NCT03750942
Title: PROphylactic Mesh to Prevent Incisional Hernias at the Former Stoma Site: the PROMISS-trial
Acronym: PROMISS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Sebastiaan van Steensel, PhD candidate, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL63259.068.17
Record Dates: First submitted 2018-11-16; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adhesix® monofilament polypropylene mesh (Bard Davol) group (Experimental): The intervention arm will receive a mesh surrounding the stoma at the time of creation of the stoma.
  Interventions: Device: Adhesix® monofilament polypropylene mesh (Bard Davol)
- Control group (No Intervention): The control group will not receive a mesh and the stoma will be created according local protocol.

INTERVENTIONS:
Device: Adhesix® monofilament polypropylene mesh (Bard Davol) — The intervention group will receive preventive mesh placement and in the control group no mesh is placed, the stoma is closed according to standard practise.
  Arms: Adhesix® monofilament polypropylene mesh (Bard Davol) group

SUMMARY:
Rationale:

Approximately 7000 stomata are created in the Netherlands every year. The occurrence of a parastomal herniation is high, with a reported incidence of 4-48%. Also, the former stoma site is at increased risk for the development of an incisional hernia. A clinical incisional hernia rate of 30% is reported after stoma reversal. Herniation can cause pain, deformity and possibly incarceration, which results in a significant impact on the quality of life of the patient.

The hypothesis of this study is that the use of a prophylactic mesh at the time of stoma formation leads to a lower incidence of incisional hernias after stoma reversal, an improved quality of life and therefore a possible cost reduction in healthcare.

Objective:

To evaluate the incidence of incisional hernias after stoma reversal after preventive mesh placement compared to no mesh placement. In addition, we aim to assess the effect of preventive mesh placement on the quality of life and the effect on healthcare cost reduction by avoiding re-intervention.

Study design:

A multicentre double blind randomized controlled trial with a total follow up of 24 months.

Study population:

Adults (18-99) undergoing bowel resection with the formation of a temporary stoma.

Intervention:

A preventive mesh will be placed using a sublay keyhole technique (pre-peritoneal, retromuscular) at stoma formation. The mesh will be left in situ after stoma reversal and the hole in the mesh will be closed, to prevent incisional herniation.

Main study parameters/endpoints:

* Primary: Incidence of incisional hernias after stoma reversal
* Secondary: Quality of life, stoma related prolapse or parastomal herniation, cost effectiveness and mesh related complications.

Nature and extent of the burden and the risks associated with participation, benefit and group relatedness:

The standard surgical procedure for the treatment of parastomal hernias is used in a prophylactic fashion. As this is standard care in parastomal hernias the risks are minimal. The mesh that is used is CE approved. The burden of participation in this study is minimal for the patient all follow-up visits coincide with the regular visits for colorectal cancer. Hence, no extra outpatient department visits, and even no additional diagnostics nor other medical procedures that could potentially burden the patient, are required.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosed with colorectal carcinoma
* Bowel resection following stoma formation, intended to be temporary.
* Elective surgery
* ASA-score I-III
* Signed informed consent

Exclusion Criteria:

* Emergency operation
* Peritonitis (i.e. bowel perforation)
* Bowel obstruction
* A life expectancy of less than 2 years (distant metastasis i.e. located in the liver, peritoneum, lung, cerebral or bone)
* Earlier hernia repair with mesh placed in a 10cm proximity of the future stoma site.
* Chronic use of antibiotics
* Chronic use of immunosuppressive medication
* ASA-score IV or above
* Not able to sign informed consent
* Patient being unable to speak Dutch
* Patient allergic to one of the components of the mesh

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of incisional hernia at the former stoma site. | 24 months
  Incidence of incisional hernia Expressed in % ranging from 0-100%, a lower percentage is considered a better outcome.

SECONDARY OUTCOMES:
Occurrence of parastomal hernia | 24 months
  Incidence of parastomal hernia Expressed in % ranging from 0-100%, a lower percentage is considered a better outcome.
Occurence of prolapse | 24 months
  Incidence of prolapse Expressed in % ranging from 0-100%, a lower percentage is considered a better outcome.
Occurence of mesh infection | 24 months
  Incidence of mesh infection Expressed in % ranging from 0-100%, a lower percentage is considered a better outcome.
Occurence of wound infections | 24 months
  Incidence of wound infections Expressed in % ranging from 0-100%, a lower percentage is considered a better outcome.
Occurence of Seroma | 24 months
  Incidence of seroma Expressed in % ranging from 0-100%, a lower percentage is considered a better outcome.
Quality of life score | 24 months
  Quality of life postoperatively assessed through questionnaires.
  - EQ-5D-5L (0-25), lower is considered a better outcome
Quality of life score | 24 months
  Quality of life postoperatively assessed through questionnaires.
  - Carolina Comfort scale (0-40), lower is considered a better outcome.
Quality of life score | 24 months
  Quality of life postoperatively assessed through questionnaires.
  - EORTC QLQ-CR29 (0-228), lower is considered a better outcome.
Operation length | during operation
  Time from start of the operation to finish (min), longer operation time can be an indication of a more complex procedure.
Time to stoma reversal | time from stoma creation to reversal
  Time between creation of the stoma and its reversal, will be expressed in days. (minimum of 14 days to a maximum of 730 days). It will be measured from creation of stoma to reversal, which is 6 weeks on average, if the stoma is not reversed within 24 months the patient is excluded. For it will not be able to reach the primary endpoint. Delay of reversal of the stoma may indicate that patient condition or other patient related factors are not optimal.
Cost-effectiveness | 24 months
  Cost benefit analysis involving health cost and societal cost due to inability to participate in work. Lower health care cost are considered a better outcome, it is hypothesised that preventive treatment results in less cost by avoiding reoperations and readmission on the long term.
  Assessment will be performed using questionnaires; the iMCQ questionnaires for cost effectiveness analysis.
  The questions of the questionnaire will be analysed separately, for the questions range from yes/no questions to multiple choice or questions regarding number of days/ hours worked.
Cost-effectiveness | 24 months
  Cost benefit analysis involving health cost and societal cost due to inability to participate in work. Lower health care cost are considered a better outcome, it is hypothesised that preventive treatment results in less cost by avoiding reoperations and readmission on the long term.
  Assessment will be performed using questionnaires; the iPCQ questionnaires for cost effectiveness analysis.
  The questions of the questionnaire will be analysed separately, for the questions range from yes/no questions to multiple choice or questions regarding number of days/ hours worked.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole D Bouvy, MD, PhD, Principal Investigator — Maastricht University Medical Centre, department of Surgery
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vu BK, Lam J, Sherman MJ, Tam MS. Prophylactic Biosynthetic Retrorectus Mesh Placement During Stoma Reversal Reduces the Rate of Stoma Site Incisional Hernia. Perm J. 2024 Jun 14;28(2):16-25. doi: 10.7812/TPP/23.115. Epub 2024 Apr 23. PMID 38652519